CLINICAL TRIAL: NCT05063175
Title: The Influences of Kyphotic Posture Correction on Balance and Risk of Fall in Children With Cerebral Palsy.
Brief Title: Correction for Kyphotic Posture for Improving Balance in Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umm Al-Qura University (Other)
Responsible Party: Principal Investigator, Ehab Mohamed Abd El Kafy, Professor of Physical Therapy, Umm Al-Qura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19-MED-01-0005
Record Dates: First submitted 2021-09-21; First posted 2021-09-30 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: Kyphosis
Keywords: Kyphosis; Balance; Fall Risk
MeSH Terms: conditions — Kyphosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Children in the control group received the conventional physical therapy protocol which was prescribed to correct the kyphotic posture of the dorsal spine, and improve postural balance stability during standing and walking.
  Interventions: Other: Conventional Physical Therapy Protocol
- Experimental Group (Experimental): The children in the experimental group received the conventional protocol applied to the control group. Further, they wore TheraTog orthotic undergarment with its strapping system for 8 hours daily for 12 successive weeks.
  Interventions: Other: Conventional Physical Therapy Protocol; Other: TheraTog orthotic undergarment with its strapping system

INTERVENTIONS:
Other: Conventional Physical Therapy Protocol — The conventional physical therapy protocol was prescribed to correct the kyphotic posture of the dorsal spine, and improve postural balance stability during standing and walking. The conventional therapeutic protocol for every child was three sessions per week for 12 successive weeks. Every treatment session was applied for two hours with a few minutes rest in between them.
Other: TheraTog orthotic undergarment with its strapping system — TheraTog orthotic undergarment with its strapping system was conducted for 8 hours daily for 12 successive weeks. It is made to be fitted directly on the skin as undergarments.
  Arms: Experimental Group

SUMMARY:
Children with spastic diplegia are at an increased risk of spinal deformities. The most common types of these spinal deformities are scoliosis and kyphosis. Thoracic hyper-kyphosis may adversely affect balance in children with cerebral palsy . The treatment approaches for hyper-kyphosis involved both conservative and surgical treatments. The Conservative approach includes corrective exercises, positioning, and spinal braces. This study aimed to evaluate the effect of conservative orthotic management for kyphotic posture on balance control, and fall risk in cerebral palsied children of spastic diplegia.

DETAILED DESCRIPTION:
Kyphosis is a posterior convexity of the spine. Children with cerebral palsy show a higher probability of progression of the kyphotic curve. If it is not adequately treated, it becomes fixed where it requires surgical management. Children with cerebral palsy have more probability to balance impairment and falls than normal children and the consequences of that fall are great. The current studies do not properly examine the effectiveness of conservative orthoses on the therapeutic management of kyphosis in children with cerebral palsy. Also, there is a shortage of studies that evaluate how correction of the thoracic kyphosis influences the balance performance and fall risk in children with cerebral palsy. TheraTogs orthosis which consists of an orthotic undergarment and external strapping system has been designed to provide a soft and passive body compression to maintain a typical body postural alignment and to improve posture control. Therefore, the objective of this study was to investigate how the correction of dorsal hyper-kyphotic posture by the TheraTogs orthotic system could influence balance control, and fall risk in cerebral palsied children of spastic diplegia.

ELIGIBILITY:
The inclusion criteria were:

* Children with a diagnosis of cerebral palsy of spastic diplegia.
* They were all between 8 and 10 years old, of both sexes.
* The degree of spasticity in the affected upper and lower extremity, was ranged between grades (1, 1+&2) according to Modified Ashworth Scale (MAS).
* Children were cognitively able to understand and follow instructions.
* The levels of their gross motor function were between level I and II according to the Gross - Motor Function Classification System (GMFCS).
* They were able to stand alone for five to ten minutes without any assistance.
* The degree of the spinal kyphosis in the sagittal plane did not exceed 45° (Cobb's angle).

The exclusion criteria were:

* Children with any orthopedic condition or fixed deformity that interfere with the spinal and limbs functions.
* Children who demonstrated allergic reactions to the adhesive tape or any other materials used in this study.
* Children with surgical interference for the lower limb and spine within the previous 2 years.
* Children with seizures, visual impairments, or perceptual problems.

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Change in the thoracic kyphosis angle (°) | [Data was collected at baseline, and 12 weeks after intervention commencement.]
  The following device (DIERS Formetric 3D/4D spine & posture analysis system) was used to examine the change in the thoracic kyphosis angle (°). This device supplies a thorough report about the alignment of the whole spine in one assessment session. It was used for assessing the sagittal plane of the back surface of the body according to a contactless 3D - scan.
Change in the thoracic flexion and extension range of motion (degree). | [Data was collected at baseline, and 12 weeks after intervention commencement.]
  Spinal mouse, a computerized spinal evaluating device, was used for evaluating the range of motion of the spinal segment in a non-invasive way. The extension and flexion range of motion of the spine were measured by the spinal mouse. The measurements were recorded from the standing position of the children.
Change in the Overall Stability Indices {percentage value (%)} for the Fall Risk Test (test that assessed the change in postural stability) | [Data was collected at baseline, and 12 weeks after intervention commencement.]
  The Biodex Balance System was used to assess the Change in the Overall Stability Index of the Fall Risk Test. In this study, the dynamic level 12 was selected for applying the fall risk test. The result for every child was registered and compared to the normative data stored in the software of the device based on children age range.
Change in the Pediatric Balance Scale score (scale that assess the change in balance performance) | [Data was collected at baseline, and 12 weeks after intervention commencement.]
  The Pediatric Balance Scale is a functional test that is used to evaluate balance impairments in children with motor deficits. The test consists of 14 tasks that assess balance performance in children. 0-4 is the rating score for each item, where zero is the minimum score and 56 is the maximum score for all tasks.

CONTACTS AND LOCATIONS:
Overall Officials: Ehab M Abd El Kafy, Ph.D, Principal Investigator — Faculty of Applied Medical Sciences - Umm Al Qura University
Locations (1):
- Umm Al Qura University, Mecca, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
- The data available is Case-by-case basis at the discretion of Primary Sponsor
Supporting Information: SAP
Time Frame: Start Date: Beginning one year following main results publication End Date: Ending two years following main results publication
Access Criteria: Data can be obtained by Principal Investigator Email Address: emkafy@uqu.edu.sa